CLINICAL TRIAL: NCT05674110
Title: Screening, Education, and Nutrition to Address Diabetes and Food Insecurity for Individuals at a Food Pantry
Brief Title: Screening and Nutrition for Patients With Diabetes: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Villanova University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2022-228
Record Dates: First submitted 2022-12-09; First posted 2023-01-06 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus
Keywords: Food Insecurity; Community Based Participatory Research; Education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education and Support (Experimental): online education and support meetings
  Interventions: Behavioral: DSMES Intervention

INTERVENTIONS:
Behavioral: DSMES Intervention — This study will provide participants with on-line education, plus weekly text messaging that will contain messages of support or encouragement sent to participants in the individual's preferred language (English or Spanish). Participants will be encouraged to attend monthly group support meetings to review the content and address any questions. Group meetings will occur at 3-time intervals (end of months: 1, 2, and 3). Group support meetings will be held in-person at a food pantry and moderated by peer mentors, nursing students, registered dietitian nutritionist (RDN), and/or a diabetes care and education specialist (DCES). Group support meetings will be held in Spanish and/or English, with no more than 10 participants in a group at one time, and will last approximately 50 minutes. For the duration of the study, participants will continue to receive monthly food items from the food pantry.

SUMMARY:
The goal of this project is to provide diabetes self-management education and support (DSMES) and simultaneously address food insecurity for a high-risk, ethnically diverse adult population who participate in a food pantry. This project will utilize a Community-Based Participatory Research model (CBPR). Community representatives will engage in project implementation by participating in designing the messaging for cultural impact and advising in study operations. This intervention targets food pantry clients self-reporting a T2DM diagnosis or who screen positive for T2DM through on-site HbA1c testing. Once enrolled, participants will complete self-paced web-based/mobile DSMES modules, available in English and Spanish, that include the ADCES7 (Association of Diabetes Care and Education Specialists) Self-Care BehaviorsTM. Support through text messaging, monthly group sessions, and peer mentorship will be facilitated by nursing students, registered dietitian nutritionists (RDNs), and diabetes care and education specialists (DCES) for 12 weeks. Participants will receive nutritious food from the pantry consistent with dietary guidelines for diabetes.

DETAILED DESCRIPTION:
Eligible patients who agree to participate in the study will be screened for diabetes via HbA1c fingerstick measurement. Participants will receive diabetes self-management education, food items recommended by registered dietitians, peer support, monthly in-person group support sessions held at the foot pantry, and text messaging with continued education. Data will be collected at intake. Follow up data will be collected 90 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Existing and/or new diagnosis of T2DM
* Food pantry participants
* English and/or Spanish speaking
* Willing/able to provide informed consent
* Must have a mobile device able to receive text messages

Exclusion Criteria:

* Under the Age of 18
* No T2DM or do not meet HbA1c > 6.5 criteria
* Not a food pantry participant
* Unwilling/unable to provide informed consent
* Spoken language is other than English/Spanish
* Individuals who do not have access to a mobile device or are unable to receive text messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes knowledge | Baseline and three months
  The Diabetes Knowledge Test (DKT2) will test change in diabetes knowledge (measured at baseline and post-intervention completion).

SECONDARY OUTCOMES:
Change in Diabetes Self-Efficacy | Baseline and three months
  Change in Diabetes self-efficacy will be measured with the Diabetes Self-Efficacy Scale which will measure individuals' perception of their ability to manage their diabetes (measured at baseline and post intervention completion).
Change in eating behaviors | Baseline and three months
  Change in eating behaviors will be measured with the Food Frequency Questionnaire (FFQ) and 3 day dietary recall at 3 months (measured at baseline and post-intervention completion).
Change in Hemoglobin A1c | Baseline and six months
  All participants will provide a fingerstick blood sample collected at 3-months following completing of the intervention. A1C is a measure of glycemic control over the last 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christina R Whitehouse, Principal Investigator — Villanova University
Locations (1):
- Villanova University, Villanova, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No